CLINICAL TRIAL: NCT06877065
Title: Role of MRI Assessment in Fertility Sparing Treatment for Cervical Cancer at Staging and Follow-up and for Identification of Risk Factors for Aggressive Disease.
Acronym: FEST-CC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6280
Record Dates: First submitted 2024-02-07; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: In the retrospective phase of the research, all patients with histological diagnosis of cervical cancer, stage FIGO up to IB2-IIA1 (T size < 4 cm), treated with fertility sparing techniques, from 2018 to 2023, will be identified retrospectively, searching on RedCap database. Of these patients, only those with good quality of MR images (available on digital support) will be selected.
- Prospective cohort: In the prospective phase of the research, all patients with histological diagnosis of cervical cancer, FIGO stage up to IB2-IIA1 (T size < 4 cm), that wish to preserve fertility and are suitable for fertility sparing treatments. Of these patients, only those with good quality of MR images (available on digital support) will be selected.

SUMMARY:
The purpose of this study is to investigate the role of MRI, including DWI, in the staging and evaluation of response to fertility sparing treatment, including both primary surgery Protocol FeST-CC V.1.0 of November 10, 2023 Pag. 5 | 23 (RT or CKC) or after NACT, followed by CKC, in patients with ECC (FIGO 2018 stage IB1- IIA1), desiring to preserve their fertility.

DETAILED DESCRIPTION:
Cervical cancer represents the fourth-most common cancer in women and the leading gynaecologic malignancies, accounting approximately 570,000 cases and 311,000 deaths in 2018 worldwide. In Europe, during last years, both mean age of pregnant women and number of nulliparous women have increased (2). Age-specific incidence data indicate that 43% of patients with cervical cancer have less than 45 years. As consequence, numerous young women diagnosed with cervical cancer are still desiring to become pregnant.

In women with early-stage cervical cancer (ECC), fertility-sparing surgery techniques include laparoscopic, abdominal or vaginal radical trachelectomy (RT) and cold knife conization (CKC) with or without pelvic lymph nodes dissection. Currently, RT is proposed as fertility-sparing surgery (FSS), alternative to radical hysterectomy, in patients with ECC staged IA1-IB1, as by the 2018 International Federation of Gynecology and Obstetrics (FIGO) classification. According to a recent metanalysis, RT and CKC present similar oncologic outcomes in terms of recurrence rates but CKC presents better obstetrical outcomes in terms of pregnancy rate (36% for CKC vs. 20% for RT) . NCCN suggested RT as an alternative to radical hysterectomy (RH) in young women desiring to preserve fertility with: disease limited to cervix, tumor size < 2 cm (or < 2.5 cm if exophytic lesion), absence of parametrial extension, an estimated distance of ≥ 1 cm from the proximal aspect of the tumor to the internal os, absence of lymphadenopathies or metastatic disease. Some authors have proposed neoadjuvant chemotherapy (NACT) followed by CKC as a safe and effective approach in ECC FIGO stage IB2.

In 2018 FIGO staging was revised allowing the use of any of the imaging modalities (i.e.

ultrasound, CT, MRI, positron emission tomography (PET)), to provide information on tumor size, nodal status, and local or systemic spread. MRI is reported to be very accurate in selecting patients eligible for FSS, in tumor size evaluation and deep stromal invasion assessment. In the evaluation of parametrial invasion, the specificity and negative predictive value of MRI were 97% and 100%, respectively.

Furthermore, MRI has demonstrated very high sensitivity and specificity in assessment of internal os involvement, 90% and 98% respectively. Moreover, MRI including diffusion-weighted imaging (DWI) assumes an important role in the evaluation of tumor response after chemotherapy. In addition, MRI is highly sensitive and accurate (90.7% and 91.7% respectively) in tumor size evaluation after FSS, especially in patients who have undergone cone biopsy before MRI examination.

The purpose of this study is to investigate the role of MRI, including DWI, in the staging and evaluation of response to fertility sparing treatment, including both primary surgery (RT or CKC) or after NACT, followed by CKC, in patients with ECC (FIGO 2018 stage IB1- IIA1), desiring to preserve their fertility.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical cancer FIGO stage up to IB2-IIA1 (T size < 4 cm) wishing to preserve fertility treated at the Oncological Gynecology Unit of Foundation Policlinico Universitario Agostino Gemelli.
* absence of nodal disease,
* no menopausal status
* wish to preserve fertility
* refusal of radical treatment.
* Patients who had a pre-treatment and post-treatment magnetic resonance imaging.
* Availability of digital MR images and histopathological samples.

Exclusion Criteria:

* Patients aged under 18 years.
* Neuroendocrine cervical tumours or other rare histology, such as glassy cells or clear cell carcinoma non-HPV related adenocarcinoma.
* ongoing pregnancy at the time of diagnosis.
* Patients without available MR images on digital media or with low quality images.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidate patients will be enrolled among those with cervical cancer, according to inclusion criteria. They will be informed about the possibility of being enrolled in this study during the outpatient clinics/hospitalization examination and will be given an adequate description of this study (objectives of the study, what the participation involves, possible risks and benefits, what the non- participation may entail, possibility of interruption, etc.). In case of enrolment, an informed consent including acceptance to make available the anonymized personal, clinical-laboratory and diagnostic imaging data will be signed.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI accuracy in preoperative staging of early stage cervical cancer for fertility-sparing treatment | 3 years
  The primary objective is to investigate the role of MRI in preoperative staging of early stage cervical cancer, in patients eligible for fertility-sparing treatment (FIGO stage up to IB2-IIA1 with T size < 4 cm).

SECONDARY OUTCOMES:
The accuracy of MRI in evaluating treatment response after fertility-sparing treatment in cervical cancer, including specificity and sensibility | 3 years
  To assess the accuracy of MRI in evaluating treatment response after fertility-sparing treatment in cervical cancer.
Assessment of MRI Parameter to predict more aggressive disease | 3 years
  To assess if MRI parameters correctly predict more aggressive disease at the time of diagnosis before fertility-sparing treatment, in correlation with the Annual Recurrence Risk Model (ARRM) both in terms of disease-free survival (DFS) and overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Benedetta Gui, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Advanced Radiology Center- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No